CLINICAL TRIAL: NCT03748706
Title: A Phase 2a, Open-label, Multiple Dose, Safety, Pharmacokinetic and Biomarker Study of PTl-125 in Mild-to-moderate Alzheimer's Disease Patients
Brief Title: PTI-125 for Mild-to-moderate Alzheimer's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: Cassava Sciences, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTI-125-03; R44AG060878 (NIH)
Record Dates: First submitted 2018-11-13; First posted 2018-11-21 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Simufilam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Simufilam (PTI-125) (Experimental): Simufilam (PTI-125) 100 mg oral tablets administered twice daily (BID)
  Interventions: Drug: PTI-125, 100 mg tablets

INTERVENTIONS:
Drug: PTI-125, 100 mg tablets — PTI-125, 100 mg tablets taken twice a day for 28 days

SUMMARY:
This is a Phase 2a, multi-center, open-label study of PTI-125 in mild-to-moderate Alzheimer's disease patients.

DETAILED DESCRIPTION:
This is a Phase 2a, multi-center, open-label study of PTI-125 in mild-to-moderate AD patients, 50-85 years of age. A total of twelve (12) patients will be enrolled into the study. Patients will receive 100 mg b.i.d. of PTI-125. The objectives of this study are to investigate the safety, pharmacokinetics and effect on biomarkers of PTI-125 following 28-day repeat-dose oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Ages >= 50 and <= 85 years
* Informed consent form (ICF) signed by the subject or legally acceptable representative.
* Clinical diagnosis of dementia due to possible or probable Alzheimer's disease
* Mini-Mental State Examination score >= 16 and <= 24 at screening
* If female, postmenopausal for at least 1 year
* Patient living at home, senior residential setting, or an institutional setting without the need for continuous (i.e. 24-hour) nursing care
* General health status acceptable for participation in the study
* Fluency (oral and written) in English or Spanish
* If receiving memantine, rivastigmine, galantamine or an AChEI, receiving a stable dose for at least 3 months (90 days) before screening and with continuous dosing for at least 3 months. If receiving donepezil, receiving any dose lower than 23 mg once daily.
* The patient is a non-smoker for at least 12 months.
* The patient or legal representative must agree to comply with the drawing of blood samples and with a lumbar puncture and the drawing of cerebrospinal fluid samples.
* The patient has a ratio of total tau/Abeta42 in cerebrospinal fluid >= 0.30.
* Patient has a caregiver or legal representative responsible for administering the drug and recording the time.

Exclusion Criteria:

* Exposure to an experimental drug, experimental biologic or experimental medical device within the longer of 5 half-lives or 3 months before screening
* Residence in a skilled nursing facility
* Clinically significant laboratory test results
* Clinically significant untreated hypothyroidism (if treated, thyroid-stimulating hormone level and thyroid supplementation dose must be stable for at least 6 months before screening)
* Insufficiently controlled diabetes mellitus or requiring insulin
* Renal insufficiency (serum creatinine >2.0 mg/dL)
* Malignant tumor within 3 years before screening (except squamous and basal cell carcinoma or cervical carcinoma in situ or localized prostate cancer or localized stage 1 bladder cancer)
* History of ischemic colitis or ischemic enterocolitis
* Unstable medical condition that is clinically significant in the judgment of the investigator
* Alanine transaminase (ALT) or aspartate transaminase (AST) >2 times the upper limit of normal or total bilirubin greater than the upper limit of normal.
* History of myocardial infarction or unstable angina within 6 months before screening
* History of more than 1 myocardial infarction within 5 years before screening
* Clinically significant cardiac arrhythmia (including atrial fibrillation), cardiomyopathy, or cardiac conduction defect (patients with a pacemaker are acceptable)
* Symptomatic hypotension, or uncontrolled hypertension
* Clinically significant abnormality on screening electrocardiogram (ECG), including but not necessarily limited to a confirmed corrected QT value >= 450 msec for males or >= 470 msec for females.
* Stroke within 18 months before screening, or history of a stroke concomitant with onset of dementia
* History of brain tumor or other clinically significant space-occupying lesion on CT or MRI
* Head trauma with clinically significant loss of consciousness within 12 months before screening or concurrent with the onset of dementia
* Onset of dementia secondary to cardiac arrest, surgery with general anesthesia, or resuscitation
* Specific degenerative CNS disease diagnosis other than Alzheimer's disease (eg, Huntington's disease, Creutzfeld-Jacob disease, Down's syndrome, Frontotemporal Dementia, Parkinson's disease)
* Wernicke's encephalopathy
* Active acute or chronic Central Nervous System infection
* Donepezil 23 mg or greater quaque die currently or within 3 months prior to enrollment in the study
* Discontinued AChEI < 30 days prior to enrollment in the study
* Antipsychotics; low doses are allowed only if given for sleep disturbances, agitation and/or aggression, and only if the subject has received a stable dose for at least 3 months before enrollment in the study
* Tricyclic antidepressants and monoamine oxidase inhibitors; all other antidepressants are allowed only if the subject has received a stable dose for at least 3 months before enrollment in the study
* Anxiolytics or sedative-hypnotics, including barbiturates (unless given in low doses for benign tremor); low doses of benzodiazepines and zolpidem are allowed only if given for insomnia/sleep disturbance, and only if the subject has received a stable dose for at least 3 months before enrollment in the study
* Peripherally acting drugs with effects on cholinergic transmission
* Immunosuppressants, including systemic corticosteroids, if taken in clinically immunosuppressive doses (Steroid use for allergy or other inflammation is permitted.)
* Antiepileptic medications if taken for control of seizures
* Chronic intake of opioid-containing analgesics
* Sedating H1 antihistamines
* Nicotine therapy (all dosage forms including a patch), varenicline (Chantix), or similar therapeutic agent within 30 days before screening
* Clinically significant illness within 30 days of enrollment
* History of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease
* Positive serum hepatitis B surface antigen (HBsAg) or positive hepatitis C virus (HCV) antibody test at screening
* Positive HIV test at screening
* Loss of a significant volume of blood (> 450 mL) within 4 weeks prior to the study
* Metformin or cimetidine.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Burns, PhD, Study Director — Cassava Sciences, Inc.
Locations (2):
- United States (2):
  - Insite Clinical Research, DeSoto, Texas
  - Clinical Trials of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang HY, Lee KC, Pei Z, Khan A, Bakshi K, Burns LH. PTI-125 binds and reverses an altered conformation of filamin A to reduce Alzheimer's disease pathogenesis. Neurobiol Aging. 2017 Jul;55:99-114. doi: 10.1016/j.neurobiolaging.2017.03.016. Epub 2017 Mar 31. PMID 28438486
- [Background] Wang HY, Bakshi K, Frankfurt M, Stucky A, Goberdhan M, Shah SM, Burns LH. Reducing amyloid-related Alzheimer's disease pathogenesis by a small molecule targeting filamin A. J Neurosci. 2012 Jul 18;32(29):9773-84. doi: 10.1523/JNEUROSCI.0354-12.2012. PMID 22815492
- [Result] Wang HY, Pei Z, Lee KC, Lopez-Brignoni E, Nikolov B, Crowley CA, Marsman MR, Barbier R, Friedmann N, Burns LH. PTI-125 Reduces Biomarkers of Alzheimer's Disease in Patients. J Prev Alzheimers Dis. 2020;7(4):256-264. doi: 10.14283/jpad.2020.6. PMID 32920628

RESULTS

PARTICIPANT FLOW:
Groups:
- PTI-125: PTI-125 100 mg oral tablets administered twice daily (BID)
  PTI-125, 100 mg tablets: PTI-125, 100 mg tablets taken twice a day for 28 days
Period: Overall Study
Arm/Group | PTI-125
Started | 13
Completed | 12
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | PTI-125
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: Years] | 67.8 [56 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Blood draws will be done to evaluate levels of PTI-125 in the plasma using non-compartmental methods in WinNonlin.
Time Frame: Study Day 1 and Day 28 at 20, 40, and 60 min and at 1.5, 2, 2.5, 3, 4, 6, 8, 10 and 12 h post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PTI-125
Number analyzed (Participants) | 13
ng/mL
  Day 1 Cmax | 1020 (442)
  Day 28 Cmax | 1100 (417)

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Levels of PTI-125 will be assessed to determine how long it takes to reach the Cmax
Time Frame: Study Day 1 and Day 28 at 20, 40, and 60 min and at 1.5, 2, 2.5, 3, 4, 6, 8, 10 and 12 h post-dose
Measure: Median (Full Range); unit: hours
Arm/Group | PTI-125
Number analyzed (Participants) | 13
hours
  Day 1 Tmax | 2.00 [1.00 to 3.00]
  Day 28 Tmax | 2.06 [1.00 to 5.93]

3. Primary Outcome: Last Quantifiable Plasma Concentration (Clast)
Description: Levels of PTI-125 will be assessed to determine the last time point where PTI-125 can be detected.
Time Frame: Study Day 1 and Day 28 at 20, 40, and 60 min and at 1.5, 2, 2.5, 3, 4, 6, 8, 10 and 12 h post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PTI-125
Number analyzed (Participants) | 13
ng/mL
  Day 1 Clast | 176 (112)
  Day 28 Clast | 238 (168)

4. Primary Outcome: Time to Last Quantifiable Plasma Concentration (Tlast)
Description: Levels of PTI-125 will be assessed to determine the elapsed time to where PTI-125 can last be detected in the plasma.
Time Frame: Study Day 1 and Day 28 at 20, 40, and 60 min and at 1.5, 2, 2.5, 3, 4, 6, 8, 10 and 12 h post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PTI-125
Number analyzed (Participants) | 13
hours
  Day 1 Tlast | 12.0 (0.0150)
  Day 28 Tlast | 12.0 (0.0285)

5. Primary Outcome: Area Under the Curve (AUClast)
Description: AUC for PTI-125 plasma concentration from time zero to the last quantifiable plasma concentration.
Time Frame: Study Day 1 and Day 28 at 20, 40, and 60 min and at 1.5, 2, 2.5, 3, 4, 6, 8, 10 and 12 h post-dose
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | PTI-125
Number analyzed (Participants) | 13
h*ng/mL
  Day 1 AUClast | 5320 (2230)
  Day 28 AUClast | 6700 (3240)

6. Primary Outcome: Plasma Half-life (T1/2)
Description: Assessment of the half-life in plasma of PTI-125
Time Frame: Study Day 1 and Day 28 at 20, 40, and 60 min and at 1.5, 2, 2.5, 3, 4, 6, 8, 10 and 12 h post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PTI-125
Number analyzed (Participants) | 13
hours
  Day 1 T1/2 | 4.51 (2.43)
  Day 28 T1/2 | 4.35 (1.39)

7. Secondary Outcome: SavaDx (Biomarker)
Description: Blood samples will be tested for the complementary diagnostic/biomarker for Alzheimer's disease.
Time Frame: Study Day 1 and Day 28
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | PTI-125
Number analyzed (Participants) | 13
% change from baseline | -39.8 (0.19)

8. Secondary Outcome: CSF Biomarkers
Description: A cerebrospinal fluid sample collection will be performed for Aβ42, tau, YKL40 and other potential CSF biomarkers
Time Frame: Change from Baseline to Day 28
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | PTI-125
Number analyzed (Participants) | 13
% change from baseline
  Total tau | -19.8 (0.04)
  Abeta42 | 4.3 (0.05)
  p-tau181 | -34.4 (0.05)
  Neurogranin | -32 (0.02)
  Neurofilament light chain | -22 (0.02)
  YKL-40 | -9 (0.01)
  IL-6 | -14 (0.01)
  IL-1 beta | -11 (0.01)
  TNF alpha | -5 (0.01)

ADVERSE EVENTS:
Time Frame: Within the 28-day treatment period.
Description: Moderate; mild; severe Serious; not serious Unlikely; likely; possibly related to drug treatment
Arm/Group | PTI-125
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 1/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTI-125 (N=13)
Fall (General disorders) | 1 (1) — Moderate severity; rated as unlikely to be related to treatment.
B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Flu (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Top enrolling PIs are included as authors on Cassava publications, but no individual PI has the right to publish alone without Cassava authorization.

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT03748706/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT03748706/SAP_002.pdf